CLINICAL TRIAL: NCT02452554
Title: A Phase 2 Study of IMGN901 (Lorvotuzumab Mertansine; NSC#: 783609) in Children With Relapsed or Refractory Wilms Tumor, Rhabdomyosarcoma, Neuroblastoma, Pleuropulmonary Blastoma, Malignant Peripheral Nerve Sheath Tumor (MPNST) and Synovial Sarcoma
Brief Title: Lorvotuzumab Mertansine in Treating Younger Patients With Relapsed or Refractory Wilms Tumor, Rhabdomyosarcoma, Neuroblastoma, Pleuropulmonary Blastoma, Malignant Peripheral Nerve Sheath Tumor, or Synovial Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVL1522; NCI-2015-00746 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ADVL1522; ADVL1522 (Other: Childrens Oncology Group); ADVL1522 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Results first posted 2019-08-29 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Pleuropulmonary Blastoma; Recurrent Malignant Peripheral Nerve Sheath Tumor; Recurrent Neuroblastoma; Recurrent Rhabdomyosarcoma; Recurrent Synovial Sarcoma; Wilms Tumor
MeSH Terms: conditions — Pleuropulmonary blastoma; Neurofibrosarcoma; Neuroblastoma; Rhabdomyosarcoma; Sarcoma, Synovial; Wilms Tumor | interventions — lorvotuzumab mertansine; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (lorvotuzumab mertansine) (Experimental): Patients receive lorvotuzumab mertansine IV over 1-1.5 hours on days 1 and 8. Treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Lorvotuzumab Mertansine; Other: Pharmacological Study

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Lorvotuzumab Mertansine — Given IV
  Other Names: Anti-Human NCAM-1 Monoclonal Antibody N901; BB-10901; huN901-DM1; IMGN901
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well lorvotuzumab mertansine works in treating younger patients with Wilms tumor, rhabdomyosarcoma, neuroblastoma, pleuropulmonary blastoma, malignant peripheral nerve sheath tumor (MPNST), or synovial sarcoma that has returned or that does not respond to treatment. Antibody-drug conjugates, such as lorvotuzumab mertansine, are created by attaching an antibody (protein used by the body?s immune system to fight foreign or diseased cells) to an anti-cancer drug. The antibody is used to recognize tumor cells so the anti-cancer drug can kill them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy of IMGN901 (lorvotuzumab mertansine) in Wilms tumor, rhabdomyosarcoma, neuroblastoma and other cluster of differentiation (CD)56-expressing tumors such as pleuropulmonary blastoma, malignant peripheral nerve sheath tumor (MPNST) and synovial sarcoma.

II. To determine the tolerability of the adult recommended phase 2 dose (RP2D) of IMGN901 administered as an intravenous infusion, administered on days 1 and 8 of a 21-day cycle, to children with refractory Wilms tumor, rhabdomyosarcoma, neuroblastoma, pleuropulmonary blastoma, MPNST, or synovial sarcoma.

III. To define and describe the toxicities of IMGN901 administered on this schedule.

EXPLORATORY OBJECTIVES:

I. To correlate tumor response with tumor CD56+ expression. II. To characterize the pharmacokinetics of IMGN901 in children with refractory cancer, including an assessment of impact on circulating CD56+ peripheral blood cells.

OUTLINE:

Patients receive lorvotuzumab mertansine intravenously (IV) over 1-1.5 hours on days 1 and 8. Treatment repeats every 21 days for up to 17 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had histologic verification of one of the malignancies listed below at original diagnosis or at relapse

  * Primary strata

    * Wilms tumor
    * Rhabdomyosarcoma
    * Neuroblastoma
  * Secondary strata: miscellaneous CD56-expressing tumors:

    * Pleuropulmonary blastoma
    * Malignant peripheral nerve sheath tumor (MPNST)
    * Synovial sarcoma
* Patients must have radiographically measurable disease (with the exception of those with neuroblastoma)

  * Measurable disease is defined as the presence of at least one lesion on magnetic resonance imaging (MRI) or computed tomography (CT) scan that can be accurately measured with the longest diameter a minimum of 10 mm in at least one dimension (CT scan slice thickness no greater than 5 mm)
  * Note: the following do not qualify as measurable disease:

    * Malignant fluid collections (e.g., ascites, pleural effusions)
    * Bone marrow infiltration except that detected by metaiodobenzylguanidine (MIBG) scan for neuroblastoma
    * Lesions only detected by nuclear medicine studies (e.g., bone, gallium or positron emission tomography [PET] scans) except as noted in patients with neuroblastoma who do not have measurable disease but have MIBG-avid evaluable disease
    * Elevated tumor markers in plasma or cerebrospinal fluid (CSF)
    * Previously radiated lesions that have not demonstrated clear progression post radiation
    * Leptomeningeal lesions that do not meet the measurements noted above
* Patients with neuroblastoma who do not have measurable disease but have MIBG-avid evaluable disease are eligible
* Patients must have a Lansky or Karnofsky performance status score of >= 50, corresponding to Eastern Cooperative Oncology Group (ECOG) categories 0, 1 or 2; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study
* Patients must have received standard treatment appropriate for their tumor type

  * Myelosuppressive chemotherapy: patients with solid tumors must not have received myelosuppressive chemotherapy within 3 weeks of enrollment onto this study (6 weeks if prior nitrosourea)
  * Hematopoietic growth factors: at least 14 days must have elapsed after receiving pegfilgrastim and least 7 days must have elapsed since the completion of therapy with a non-pegylated growth factor
  * Biologic (anti-neoplastic agent): at least 7 days must have elapsed since completion of therapy with a biologic agent; for agents that have known adverse events occurring beyond 7 days after administration, this period prior to enrollment must be extended beyond the time during which adverse events are known to occur
  * Monoclonal antibodies: at least 3 half-lives must have elapsed since prior therapy that included a monoclonal antibody
  * Radiotherapy: >= 2 weeks must have elapsed since local palliative external beam radiation therapy (XRT) (small port); >= 6 weeks must have elapsed since treatment with therapeutic doses of MIBG; >= 3 months must have elapsed if prior craniospinal XRT was received, if >= 50% of the pelvis was irradiated, or if total body irradiation (TBI) was received; >= 6 weeks must have elapsed if other substantial bone marrow irradiation was given
  * Stem cell transplant or rescue without TBI: no evidence of active graft vs. host disease and >= 2 months must have elapsed since transplant
* For patients with solid tumors without bone marrow involvement: peripheral absolute neutrophil count (ANC) >= 1000/uL
* For patients with solid tumors without bone marrow involvement: platelet count >= 100,000/uL (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to enrollment)
* For patients with solid tumors and known bone marrow metastatic disease: peripheral absolute neutrophil count (ANC) >= 750/uL
* For patients with solid tumors and known bone marrow metastatic disease: platelet count >= 75,000/uL (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * Age 1 to < 2 years: maximum serum creatinine: 0.6 mg/dL in males and females
  * Age 2 to < 6 years: maximum serum creatinine: 0.8 mg/dL in males and females
  * Age 6 to < 10 years: maximum serum creatinine: 1 mg/dL in males and females
  * Age 10 to < 13 years: maximum serum creatinine: 1.2 mg/dL in males and females
  * Age 13 to < 16 years: maximum serum creatinine: 1.5 mg/dL in males and 1.4 mg/dL in females
  * Age >= 16 years: maximum serum creatinine: 1.7 mg/dL in males and 1.4 mg/dL in females
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 110 U/L (for the purpose of this study, the ULN for SGPT is 45 U/L)
* Serum albumin >= 2 g/dL
* Shortening fraction of >= 27% by echocardiogram, or ejection fraction of >= 50% by gated radionuclide study
* Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Patients who are pregnant or breast-feeding are not eligible for this study; negative pregnancy tests must be obtained in girls who are post-menarchal; males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for the duration of study therapy and for 4 weeks after the last dose of study therapy; breastfeeding women are excluded
* Concomitant medications

  * Corticosteroids: patients requiring corticosteroids who have not been on a stable or decreasing dose of corticosteroid for the 7 days prior to enrollment are not eligible
  * Patients who have received previous treatment with IMGN901 are not eligible
  * Investigational drugs: patients who are currently receiving another investigational drug are not eligible
  * Anti-cancer agents: patients who are currently receiving other anti-cancer agents are not eligible
  * Anti-graft-versus-host disease (GVHD) or agents to prevent organ rejection post-transplant: patients who are receiving cyclosporine, tacrolimus or other agents to prevent either graft-versus-host disease post bone marrow transplant or organ rejection post-transplant are not eligible for this trial
* Patients who have a CNS toxicity > grade 2 are not eligible
* Patients must not have known active central nervous system (CNS) metastases; patients with known central nervous system metastases are excluded unless treated surgically or with radiotherapy, and stable with no recurrent lesions for at least 6 months
* Patients who have baseline peripheral neuropathy >= grade 2 are not eligible
* Patients who have an uncontrolled infection are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible

Ages: 12 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2015-10-12 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James I Geller, Principal Investigator — Children's Oncology Group
Locations (69):
- United States (69):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Each of 6 disease strata enrolled up to 16 patients who were evaluable for the primary response criteria.
Groups:
- Stratum 1: Wims Tumor; Stratum 2: Rhabdomyosarcoma; Stratum 3: Neuroblastoma; Stratum 4: Pleuropulmonary Blastoma; Stratum 5: Malignant Peripheral Nerve Sheath Tumor; Stratum 6: Synovial Sarcoma: ADVL1522 Dose Level 1: IMGN901 110 mg/m2/IV over 1-1.5 hours on Days 1 and 8 every 21 days, repeatable up to 17 cycles
Period: Overall Study
Arm/Group | Stratum 1: Wims Tumor | Stratum 2: Rhabdomyosarcoma | Stratum 3: Neuroblastoma | Stratum 4: Pleuropulmonary Blastoma | Stratum 5: Malignant Peripheral Nerve Sheath Tumor | Stratum 6: Synovial Sarcoma
Started | 17 | 17 | 12 | 1 | 5 | 10
Completed | 0 | 0 | 1 | 0 | 0 | 1
Not Completed | 17 | 17 | 11 | 1 | 5 | 9
Not completed — Death | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 13 | 14 | 9 | 1 | 5 | 8
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 0 | 0 | 1
Not completed — Ineligible | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Never Received Treatment | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1: Wims Tumor | Stratum 2: Rhabdomyosarcoma | Stratum 3: Neuroblastoma | Stratum 4: Pleuropulmonary Blastoma | Stratum 5: Malignant Peripheral Nerve Sheath Tumor | Stratum 6: Synovial Sarcoma | Total
Number analyzed (Participants) | 17 | 17 | 12 | 1 | 5 | 10 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 7 | 12 | 1 | 5 | 6 | 44
  Between 18 and 65 years | 4 | 10 | 0 | 0 | 0 | 4 | 18
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.61 (6.48) | 18.43 (5.28) | 7.78 (1.94) | 3.69 (NA) — There was only one participant in stratum 4, therefore a Standard Deviation can't be calculated. | 12.96 (4.29) | 17.37 (4.59) | 13.2 (6.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 3 | 1 | 4 | 6 | 27
  Male | 12 | 9 | 9 | 0 | 1 | 4 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 1 | 0 | 1 | 1 | 8
  Not Hispanic or Latino | 13 | 14 | 10 | 1 | 4 | 9 | 51
  Unknown or Not Reported | 2 | 0 | 1 | 0 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 1 | 0 | 1 | 2 | 9
  White | 10 | 14 | 10 | 1 | 3 | 5 | 43
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 1 | 0 | 0 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Objective Response by Response Evaluation Criteria in Solid Tumors Version 1.1
Description: The best response of disease will be examined separately in each stratum. A responder is defined as a patient who achieves a best response of partial response or complete response on the study. Response rates will be calculated as the percent of evaluable patients who are responders, and Clopper-Pearson confidence intervals will be constructed.
Time Frame: Up to 18 weeks (6 courses)
Population: 2 participants were excluded from analysis; 1 participant never received treatment and 1 participant was ineligible, also never receiving treatment.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Stratum 1: Wims Tumor | Stratum 2: Rhabdomyosarcoma | Stratum 3: Neuroblastoma | Stratum 4: Pleuropulmonary Blastoma | Stratum 5: Malignant Peripheral Nerve Sheath Tumor | Stratum 6: Synovial Sarcoma
Number analyzed (Participants) | 16 | 16 | 12 | 1 | 5 | 10
Percent of participants | 0.00 [0.00 to 20.59] | 6.25 [0.16 to 30.23] | 0.00 [0.00 to 26.46] | 0.00 [0.00 to 97.50] | 0.00 [0.00 to 52.18] | 0.00 [0.00 to 30.85]

2. Primary Outcome: Incidence of Toxicities of Lorvotuzumab Mertansine, Using the NCI Common Terminology Criteria for Adverse Events Version 4.0
Description: Toxicity tables will be constructed to summarize the observed incidence by type of toxicity and grade for toxicities with Possible, Probable, or Definite attribution to the study drug. Tables will summarize incidence by cycle.
Time Frame: Up to 12 months (17 courses)
Population: 203 treatment-cycles were reported for the analysis. 2 participants were excluded from analysis;1 participant never received treatment and 1 participant was ineligible, also never receiving treatment.
Measure: Number; unit: Treatment cycles
Units Other Than Participants: Treatment Cycles
Arm/Group | Treatment (Lorvotuzumab Mertansine)
Number analyzed (Participants) | 60
Number analyzed (Treatment Cycles) | 203
Treatment cycles
  Anemia: Grade 2 | 0
  Anemia: Grade 3 | 2
  Anemia: Grade 4 | 0
  Anemia: Grade 5 | 0
  Colonic fistula: Grade 2 | 0
  Colonic fistula: Grade 3 | 0
  Colonic fistula: Grade 4 | 1
  Colonic fistula: Grade 5 | 0
  Colonic perforation: Grade 2 | 0
  Colonic perforation: Grade 3 | 0
  Colonic perforation: Grade 4 | 0
  Colonic perforation: Grade 5 | 1
  Dental caries: Grade 2 | 0
  Dental caries: Grade 3 | 1
  Dental caries: Grade 4 | 0
  Dental caries: Grade 5 | 0
  Nausea: Grade 2 | 0
  Nausea: Grade 3 | 1
  Nausea: Grade 4 | 0
  Nausea: Grade 5 | 0
  Vomiting: Grade 2 | 1
  Vomiting: Grade 3 | 1
  Vomiting: Grade 4 | 0
  Vomiting: Grade 5 | 0
  Tooth infection: Grade 2 | 0
  Tooth infection: Grade 3 | 1
  Tooth infection: Grade 4 | 0
  Tooth infection: Grade 5 | 0
  Alanine aminotransferase increased: Grade 2 | 0
  Alanine aminotransferase increased: Grade 3 | 3
  Alanine aminotransferase increased: Grade 4 | 0
  Alanine aminotransferase increased: Grade 5 | 0
  Aspartate aminotransferase increased: Grade 2 | 0
  Aspartate aminotransferase increased: Grade 3 | 1
  Aspartate aminotransferase increased: Grade 4 | 0
  Aspartate aminotransferase increased: Grade 5 | 0
  Lymphocyte count decreased: Grade 2 | 0
  Lymphocyte count decreased: Grade 3 | 2
  Lymphocyte count decreased: Grade 4 | 0
  Lymphocyte count decreased: Grade 5 | 0
  Hyperglycemia: Grade 2 | 0
  Hyperglycemia: Grade 3 | 1
  Hyperglycemia: Grade 4 | 0
  Hyperglycemia: Grade 5 | 0
  Hyperuricemia: Grade 2 | 0
  Hyperuricemia: Grade 3 | 1
  Hyperuricemia: Grade 4 | 0
  Hyperuricemia: Grade 5 | 0
  Hypokalemia: Grade 2 | 0
  Hypokalemia: Grade 3 | 1
  Hypokalemia: Grade 4 | 0
  Hypokalemia: Grade 5 | 0
  Hypophosphatemia: Grade 2 | 0
  Hypophosphatemia: Grade 3 | 1
  Hypophosphatemia: Grade 4 | 0
  Hypophosphatemia: Grade 5 | 0
  Headache: Grade 2 | 1
  Headache: Grade 3 | 0
  Headache: Grade 4 | 0
  Headache: Grade 5 | 0
  Peripheral motor neuropathy: Grade 2 | 0
  Peripheral motor neuropathy: Grade 3 | 1
  Peripheral motor neuropathy: Grade 4 | 0
  Peripheral motor neuropathy: Grade 5 | 0
  Peripheral sensory neuropathy: Grade 2 | 0
  Peripheral sensory neuropathy: Grade 3 | 1
  Peripheral sensory neuropathy: Grade 4 | 0
  Peripheral sensory neuropathy: Grade 5 | 0
  All Reportable AEs: Grade 2 | 2
  All Reportable AEs: Grade 3 | 18
  All Reportable AEs: Grade 4 | 1
  All Reportable AEs: Grade 5 | 1

3. Other Pre Specified Outcome: Pharmacokinetic (PK) Parameters of Lorvotuzumab Mertansine
Description: A descriptive analysis of PK parameters of lorvotuzumab mertansine will be performed to define systemic exposure, drug clearance, and other pharmacokinetic parameters. The PK parameters will be summarized with simple summary statistics, including means, medians, ranges, and standard deviations (if numbers and distribution permit). Analyses will be descriptive and exploratory and hypotheses generating in nature.
Time Frame: Pre-treatment, end of infusion, and 2, 6, 24, 48, and 96 hours after end of infusion on day 1 of course 1, and pre-treatment, end of infusion, and 2 and 6 hours after end of infusion on day 8 of course 1
Reporting Status: Not Posted

4. Other Pre Specified Outcome: CD56 Expression
Description: The association between CD56+ expression and response will be evaluated using the exact conditional test of proportions (Fisher?s Exact test). Analyses will be descriptive and exploratory and hypotheses generating in nature.
Time Frame: Day 1 and 8 of course 1 prior to lorvotuzumab mertansine
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: While patients were on Protocol Therapy: Up to 17, 28-day cycles
Description: AE reporting is collected routinely using case report forms. The SAE table reflects NCI CTCAEs submitted by the institution, via expedited reporting (NCI AdEERs/CAeRs). The "AE Other" table reflects all CTCAEs collected; excludes those reported as SAEs. Patients who did not receive treatment before being take off study were not included in the AE tables; per protocol, AE data was not collected for those patients. Ineligible patients were excluded from both the AE and All-Cause Mortality tables.
Arm/Group | Stratum 1: Wims Tumor | Stratum 2: Rhabdomyosarcoma | Stratum 3: Neuroblastoma | Stratum 4: Pleuropulmonary Blastoma | Stratum 5: Malignant Peripheral Nerve Sheath Tumor | Stratum 6: Synovial Sarcoma
All-Cause Mortality (participants affected / at risk) | 10/17 | 11/16 | 4/12 | 1/1 | 1/5 | 2/10
Serious Adverse Events (participants affected / at risk) | 7/16 | 8/16 | 1/12 | 0/1 | 0/5 | 3/10
Other Adverse Events (participants affected / at risk) | 5/16 | 4/16 | 4/12 | 1/1 | 1/5 | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1: Wims Tumor (N=16) | Stratum 2: Rhabdomyosarcoma (N=16) | Stratum 3: Neuroblastoma (N=12) | Stratum 4: Pleuropulmonary Blastoma (N=1) | Stratum 5: Malignant Peripheral Nerve Sheath Tumor (N=5) | Stratum 6: Synovial Sarcoma (N=10)
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Colonic fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Colonic perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Death NOS (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 2
Tooth infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Optic nerve disorder (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1: Wims Tumor (N=16) | Stratum 2: Rhabdomyosarcoma (N=16) | Stratum 3: Neuroblastoma (N=12) | Stratum 4: Pleuropulmonary Blastoma (N=1) | Stratum 5: Malignant Peripheral Nerve Sheath Tumor (N=5) | Stratum 6: Synovial Sarcoma (N=10)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fever (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Irregular menstruation (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 3 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Weight loss (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT02452554/Prot_SAP_000.pdf